CLINICAL TRIAL: NCT07087652
Title: Onco Move - Improvement of Psychophysical Fitness in Adult Cancer Survivors
Acronym: OncoMove
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gdansk University of Physical Education and Sport (Other)
Collaborators: University of Cadiz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AWFiS/2025_1_MW-P
Record Dates: First submitted 2025-06-24; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-04

CONDITIONS: Cancer
Keywords: cancer exercise; oncology exercise; physical activity and cancer
MeSH Terms: conditions — Neoplasms; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The intervention group will participate in a multicomponent face-to-face Onco Move exercise training programme for 16 weeks. The intervention will include three training sessions per week (each lasting 60 minutes), held in the fitness rooms and the gym at Gdansk University of Physical Education and Sport in Poland. The intervention will include aerobic and strength exercises but also coordination/balance and flexibility, with warm-up and cool-down elements. The assessments will be conducted at four points: before the intervention, after 8 weeks, after 16 weeks, and 3 months after the intervention.
  Interventions: Other: Onco Move multicomponent face-to-face training program
- Control Group (No Intervention): The control group will not participate in the exercise training intervention during the course of the project. However, it will take part in all the assessments just like the experimental group: before the intervention, after 8 weeks, after 16 weeks, and 3 months after the intervention. The control group will be allowed to participate in the training intervention after the Onco Move project has ended.

INTERVENTIONS:
Other: Onco Move multicomponent face-to-face training program — The Onco Move intervention will include three training sessions per week (each lasting 60 minutes), held in the fitness rooms and the gym at Gdansk University of Physical Education and Sport in Poland for 16 weeks. The intervention will include aerobic and strength exercises but also coordination/balance and flexibility, with warm-up and cool-down elements.
  Arms: Intervention Group

SUMMARY:
The Onco Move project aims to assess the impact of a 16-week supervised multicomponent group exercise training program on the psychophysical well-being of individuals undergoing or recovering from cancer treatment. A total of 70 participants, aged 18-55, with various types of cancer, will be recruited for the study. Participants will be randomly assigned to either an experimental group (which will engage in the Onco Move exercise program) or a control group (usual care). Baseline measurements will be taken to assess their psychological, physiological, functional, and biochemical health. These tests will help determine the initial psychophysical health levels and the quality of life of the participants.The experimental group will undergo group exercise sessions three times a week at the Gdansk University of Physical Education and Sport, led by certified fitness instructors. The study will assess the effects of the program at three different time points: after 8 weeks, after 16 weeks, and 3 months after the completion of the program. The main objective is to investigate how regular Onco Move training influences the physical and psychological health of cancer patients, including their overall functional status, fitness, and quality of life.The findings will provide valuable insights into the positive psychophysical effects of group exercise training for cancer patients and contribute to developing a set of recommended physical activity and exercise forms for oncology patients during and after treatment. Additionally, the results will help in the creation of guidelines for recommending psychophysical exercises that could aid recovery and improve the quality of life for cancer patients.

DETAILED DESCRIPTION:
The Onco Move Project is designed to assess the effects of a 16-week supervised group exercise multicomponent program on the psychophysical well-being of individuals undergoing or recovering from cancer treatment. The study will involve 70 participants aged between 18 and 55 years, representing a diverse sample with different cancer types. The participants will be randomly assigned to one of two arms: the experimental group, which will participate in the Onco Move exercise program, or the control group, which will not engage in the exercise intervention. The primary objective of the study is to investigate how regular participation in the Onco Move exercise program affects various aspects of the participants' physical and psychological health. These aspects include overall functional status, fitness levels, and quality of life. The study will assess the impact of the training on multiple parameters, such as psychological health (e.g., anxiety, depression, and stress), physical function or health-related fitness (e.g., muscular strength, cardiorespiratory fitness, balance and body composition), autonomy (e.g., ability to perform daily activities) and biomarkers associated with inflammation, muscle recovery, and overall metabolic function, as well as genetic markers, which will help evaluate individual variability in response to the intervention and provide insights into genetic influences on inflammation, metabolism, muscle adaptation, and cellular aging.

By examining these outcomes, the study aims to provide new insights into how structured physical exercise can benefit cancer patients during and after treatment. This information could serve as the foundation for developing guidelines for recommending specific exercise programs tailored to oncology patients' needs. A total of 70 participants will be recruited for the study. Participants will be carefully selected to include individuals between the ages of 18 and 55 who have undergone or are currently undergoing cancer treatment. They will represent a variety of cancer types to ensure that the findings are applicable across different patient populations. Prior to participation, baseline measurements will be conducted to assess their psychological, physiological, functional, and biochemical health status.After the baseline assessment, participants will be randomly assigned to one of two arm: 1) Experimental group: This group will participate in the Onco Move exercise program, which involves supervised group exercise sessions held three times per week. 2) Control group: Participants in the control group will not engage in the Onco Move program but will continue their usual activities/care and they will get physical activity recommendations. They will receive general wellness advice and physical activity recommendations but will not be prescribed any specific physical exercise training during the study period.

The Onco Move exercise program is specifically designed for cancer patients and will include a combination of aerobic, strength, flexibility, and coordination/balance exercises. The exercise training sessions will be adapted to participants' individual fitness levels and will progress in load/intensity throughout the 16 weeks. The program aims to: (1) Improve aerobic capacity and muscular strength; (2) Enhance flexibility, coordination/balance, and mobility; (3) Reduce fatigue and improve mood; (4) Promote a sense of empowerment and increase overall physical activity levels. Sessions will be held three times a week, with each session lasting approximately 60 minutes (volume parameter). The exercise program will be personalized and tailored to the needs and abilities of each participant, ensuring that they engage in safe and effective exercises that are suitable for their current level of function. All sessions will be supervised by certified fitness instructors who are trained to work with individuals recovering from cancer treatment.

The impact of the Onco Move program will be evaluated at four time points during the study: (1) At the baseline; (2) After 8 weeks of participation in the exercise program; (3) After 16 weeks, at the completion of the exercise program; and (4) Three months after the completion of the program, to assess the longer-term effects of the intervention. At each time point, participants will undergo a comprehensive evaluation, including psychological, physiological, and functional assessments, as well as biochemical testing to measure specific health markers. These time points will help determine the immediate and sustained effects of the fitness program on participants' well-being.The study will use a variety of outcome measures to assess the impact of the Onco Move program. These include: (1) Physical fitness tests: A series of tests designed to assess strength, balance, flexibility, and cardiorespiratory fitness, including the Senior Fitness Test (SFT) and Short Physical Performance Battery (SPPB); (2) Psychological assessments as tools to assess anxiety, depression, stress, and quality of life, such as the Four-Item Patient Health Questionnaire For Anxiety And Depression (PHQ-4) and various scales measuring mood, sexual function, and general health-related quality of life; (3) Biochemical markers, blood samples will be analyzed to measure biomarkers such as IL-6, IL-15, Irisin, BDNF, SPARC, and decorin, which are associated with inflammation, muscle health, and overall physical recovery; (4) Genetic analyses will include polymorphisms located in the following genes: ACE, ACTN3, PPARGC1A, BDNF, VEGF, IL6, NOS3, HIF1A, TNF-α, mTOR pathway, telomeres, and telomerase; (5)Self-Reported Fitness: Participants' subjective assessments of their fitness will be recorded using tools such as the International Fitness Scale (IFIS).

The Onco Move project has the potential to make significant contributions to the field of cancer exercise research. By investigating the psychophysical effects of physical exercise training, the study will provide evidence-based insights into the benefits of structured physical exercise for cancer patients. These findings could lead to the development of guidelines for oncology professionals, helping them to recommend appropriate physical exercise during and after treatment. Furthermore, the study will help shape future exercise programs and improve quality of life for cancer survivors by promoting physical exercise as a central component of post-treatment recovery.The results of this study may also pave the way for health policy changes that encourage the integration of exercise interventions into standard cancer care practices, improving outcomes and empowering cancer survivors to take control of their physical and psychological health. By carefully assessing the effects of the Onco-Move program on various health parameters, the study aims to contribute valuable evidence that will guide the development of personalized and tailored physical exercise interventions for cancer patients. Ultimately, the project seeks to enhance the overall well-being of cancer patients and survivors, improve their quality of life, and provide a foundation for future exercise interventions in oncology care.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 55.
* Currently undergoing cancer treatment or up to 5 years post-treatment.
* Individuals with various types of cancer.
* Participants who have been physically inactive and have led a sedentary lifestyle since diagnosis.
* Both genders, with no requirement for equal distribution between women and men.
* Participants who commit to attending three training sessions per week.
* Oncologist's approval for participation in the project.
* Signed informed consent from the patient to participate in the study and consent for personal data processing.

Exclusion Criteria:

* Age below 18 or above 55 at the time of registration for the project.
* Physically active individuals.
* Health conditions preventing continued participation in the study or intervention.
* Participants who do not commit to attending three training sessions per week.
* Lack of oncologist's approval for participation in the study and training activities outlined in the project.
* Lack of signed informed consent for participation in the study and consent for personal data processing.
* Pregnant women*.

  * Pregnant women who wish to participate in the project will be allowed to attend a free lecture on the guidelines from the World Health Organization and the American College of Sports Medicine regarding recommended physical activity for cancer patients.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Assessed changes from baseline Health-Related Quality of Life (HRQOL) | From enrolment to 3 months after the intervention
  HRQOL will be assessed pre-, post-intervention, and at follow-up using validated questionnaire: European Organisation for Research and Treatment of Cancer Core Quality of Life questionnaire-Core 30 (EORTC QLQ-C30).
  This instrument measures general quality of life and includes multiple subscales (e.g. physical, emotional, cognitive functioning). Scores on each scale range from 0 to 100.
  * For functional scales and global health status, higher scores indicate better functioning or QoL.
  * For symptom scales/items, higher scores indicate more severe symptoms (i.e. worse outcomes).
  Data will be collected via digital or paper formats and analyzed. Statistical methods include repeated measures ANOVA and linear mixed-effects models to detect changes over time. Missing data will be handled via multiple imputation. This approach provides a comprehensive assessment of psychological and functional well-being related to the intervention.

SECONDARY OUTCOMES:
Change in female sexual function, assessed by Female Sexual Function Index (FSFI) | From enrolment to 3 months after the intervention
  The FSFI is a 19-item validated questionnaire measuring female sexual function across six domains: desire, arousal, lubrication, orgasm, satisfaction, and pain. Scores range from 2 to 36, with higher scores indicating better sexual function.
  Data collected via digital or paper formats will be analyzed using repeated measures ANOVA and linear mixed-effects models to assess changes over time. Missing data will be addressed with multiple imputation.
Change in male sexual function, assessed by International Index of Erectile Function (IIEF) | From enrolment to 3 months after the intervention
  The IIEF is a 15-item questionnaire assessing male sexual function, including erectile function, orgasmic function, sexual desire, intercourse satisfaction, and overall satisfaction. Scores range from 5 to 75, with higher scores indicating better sexual function. Data collected via digital or paper formats will be analyzed using repeated measures ANOVA and linear mixed-effects models to assess changes over time. Missing data will be addressed with multiple imputation.
Change in mood states, assessed by UWIST Mood Adjective Checklist (UMACL) | From enrolment to 3 months after the intervention
  UMACL measures three mood dimensions: tense arousal, energetic arousal, and hedonic tone. Scores vary by subscale; higher scores indicate greater presence of the respective mood state. Data collected via digital or paper formats will be analyzed using repeated measures ANOVA and linear mixed-effects models to assess changes over time. Missing data will be addressed with multiple imputation.
Change in perceived stress, assessed by The Feeling of Stress Questionnaire (KPS) | From enrolment to 3 months after the intervention
  KPS assesses perceived psychosocial stress across domains such as work and emotional strain. Scores vary by domain; higher scores indicate greater perceived stress. Data collected via digital or paper formats will be analyzed using repeated measures ANOVA and linear mixed-effects models to assess changes over time. Missing data will be addressed with multiple imputation.
Change in anxiety and depression symptoms, assessed by the Four-Item Patient Health Questionnaire For Anxiety And Depression (PHQ-4) | From enrolment to 3 months after the intervention
  PHQ-4 is a 4-item screening tool with two items each for anxiety and depression. Scores range from 0 to 12, with higher scores indicating more severe symptoms.
  Data collected via digital or paper formats will be analyzed using repeated measures ANOVA and linear mixed-effects models to assess changes over time. Missing data will be addressed with multiple imputation.
Change in personality traits, assessed by NEO Five-Factor Inventory (NEO-FFI) | From enrolment to 3 months after the intervention
  NEO-FFI assesses five personality traits: Neuroticism, Extraversion, Openness, Agreeableness, and Conscientiousness. Each trait is scored separately; higher scores indicate stronger presence of the trait. Data collected via digital or paper formats will be analyzed using repeated measures ANOVA and linear mixed-effects models to assess changes over time. Missing data will be addressed with multiple imputation.
Change in state and trait anxiety, assessed by State-Trait Anxiety Inventory (STAI) | From enrolment to 3 months after the intervention
  STAI includes two 20-item subscales measuring state anxiety (temporary) and trait anxiety (long-term). Scores range from 20 to 80 per subscale, with higher scores indicating greater anxiety. Data collected via digital or paper formats will be analyzed using repeated measures ANOVA and linear mixed-effects models to assess changes over time. Missing data will be addressed with multiple imputation.
Change in lower limb strength, assessed by Chair Stand Test (from Short Physical Performance Battery and Senior Fitness Test) | From enrolment to 3 months after the intervention
  Lower limb strength will be measured using the Chair Stand Test, included in both the Short Physical Performance Battery (SPPB) and the Senior Fitness Test (SFT). Participants are asked to rise from a chair without using their arms, either completing five repetitions as fast as possible (SPPB) or as many repetitions as possible in 30 seconds (SFT). Higher scores indicate better lower body strength and functional independence. Data collected via digital or paper formats will be analyzed using repeated measures ANOVA and linear mixed-effects models to assess changes over time. Missing data will be addressed with multiple imputation.
Change in upper limb strength, assessed by Arm Curl Test (from SFT) | From enrolment to 3 months after the intervention
  Upper limb strength will be assessed using the Arm Curl Test from the SFT. Participants perform as many bicep curls as possible in 30 seconds using standardized weights (2.3 kg for women and 3.6 kg for men). The number of repetitions is recorded. Higher scores indicate greater upper body muscular strength.
  Data collected via digital or paper formats will be analyzed using repeated measures ANOVA and linear mixed-effects models to assess changes over time. Missing data will be addressed with multiple imputation.
Change in flexibility, assessed by Toe Touch and Back Scratch Tests (from SFT) | From enrolment to 3 months after the intervention
  Flexibility will be assessed using two tests from the Senior Fitness Test (SFT):
  * The Toe Touch (Sit-and-Reach) Test measures lower body flexibility.
  * The Back Scratch Test measures upper body (shoulder) flexibility. Reach distances are recorded in centimeters, with positive values indicating the participant reaches beyond the target point. Higher values indicate greater flexibility.
  Data collected via digital or paper formats will be analyzed using repeated measures ANOVA and linear mixed-effects models to assess changes over time. Missing data will be addressed with multiple imputation.
Change in aerobic capacity, assessed by 6-Minute Walk or 2-Minute Step Test (from SFT) | From enrolment to 3 months after the intervention
  Aerobic capacity will be assessed using one of the two tests from the Senior Fitness Test (SFT), selected based on the participant's fitness level:
  * The 6-Minute Walk Test records the total distance walked in meters.
  * The 2-Minute Step Test counts the number of knee lifts within 2 minutes. Both tests assess cardiovascular endurance. Higher values represent better aerobic capacity.
  Data collected via digital or paper formats will be analyzed using repeated measures ANOVA and linear mixed-effects models to assess changes over time. Missing data will be addressed with multiple imputation.
Change in balance and agility, assessed by 8-Foot Up-and-Go Test (from SF) | From enrolment to 3 months after the intervention
  Balance and agility will be assessed using the 8-Foot Up-and-Go Test from the Senior Fitness Test (SFT). Participants stand up from a seated position, walk 8 feet (2.44 m), turn, return, and sit down. The time to complete the task is recorded in seconds. Lower times indicate better balance, agility, and risk reduction for falls.
  Data collected via digital or paper formats will be analyzed using repeated measures ANOVA and linear mixed-effects models to assess changes over time. Missing data will be addressed with multiple imputation.
Change in balance, assessed by Standing Balance Test (from SPPB) | From enrolment to 3 months after the intervention
  Static balance will be assessed using the Standing Balance Test from SPPB. Participants are asked to maintain three progressively more challenging foot positions (side-by-side, semi-tandem, tandem) for up to 10 seconds each. The total score ranges from 0 to 4, with higher scores indicating better balance and lower fall risk.
  Data collected via digital or paper formats will be analyzed using repeated measures ANOVA and linear mixed-effects models to assess changes over time. Missing data will be addressed with multiple imputation.
Change in walking speed, assessed by 4-Meter Walk Test (from SPPB) | From enrolment to 3 months after the intervention
  Walking speed will be assessed using the 4-Meter Walk Test from SPPB. Participants walk 4 meters at their usual pace. Time is recorded and speed is calculated in meters per second. Higher speeds indicate better physical function and are associated with reduced fall risk and improved health outcomes.
  Data collected via digital or paper formats will be analyzed using repeated measures ANOVA and linear mixed-effects models to assess changes over time. Missing data will be addressed with multiple imputation.
Change in pain threshold, assessed by AlgoMed Algometer | From enrolment to 3 months after the intervention
  Pain threshold will be evaluated at baseline, post-intervention, and follow-up using using the AlgoMed algometer, which applies calibrated pressure stimuli to assess the minimum pressure at which pain is perceived. Higher thresholds indicate lower pain sensitivity.
  Data will be analyzed using repeated measures statistical models to detect changes over time. This multimodal assessment captures both sensory and experiential aspects of pain, providing a comprehensive profile of pain sensitivity and adaptation to the intervention.
Change in pain tolerance, assessed by AlgoMed Algometer | From enrolment to 3 months after the intervention
  Pain tolerance will be measured using the AlgoMed algometer, defined as the maximum pressure tolerated before pain becomes intolerable. Higher tolerance values indicate better pain endurance. Measurements will be taken at baseline, post-intervention, and follow-up.
  Data will be analyzed using repeated measures statistical models to detect changes over time. This multimodal assessment captures both sensory and experiential aspects of pain, providing a comprehensive profile of pain sensitivity and adaptation to the intervention.
Change in subjective pain intensity, assessed by Visual Analogue Scale (VAS) | From enrolment to 3 months after the intervention
  Subjective pain intensity will be rated by participants using the Visual Analogue Scale (VAS), a 100-mm horizontal line where 0 indicates "no pain" and 100 indicates "worst imaginable pain." Higher scores indicate greater pain intensity. Assessments will occur at baseline, post-intervention, and follow-up.
  Data will be analyzed using repeated measures statistical models to detect changes over time. This multimodal assessment captures both sensory and experiential aspects of pain, providing a comprehensive profile of pain sensitivity and adaptation to the intervention.
Change in pain characteristics, assessed by Laitinen Pain Scale | From enrolment to 3 months after the intervention
  Pain characteristics will be assessed using the Laitinen Pain Scale, which evaluates four dimensions: pain intensity, frequency, use of analgesics, and limitations in physical activity. Participants rate each dimension on a scale from 0 to 4, with higher scores indicating greater severity or frequency. The total score is the sum of these four ratings, with a maximum possible score of 16. Assessments will occur at baseline, post-intervention, and follow-up.
  Data will be analyzed using repeated measures statistical models to detect changes over time. This multimodal assessment captures both sensory and experiential aspects of pain, providing a comprehensive profile of pain sensitivity and adaptation to the intervention.
Change in body weight, assessed by InBody 720 Bioimpedance Analyzer | From enrolment to 3 months after the intervention
  Body weight will be measured using a bioimpedance analyzer (InBody 720). Units: Kilograms (kg)
Change in body fat percentage, assessed by InBody 720 Bioimpedance Analyzer | From enrolment to 3 months after the intervention
  Body fat percentage will be measured using the InBody 720 bioimpedance analyzer, which estimates the proportion of fat mass relative to total body weight. Measurements will be taken at baseline, post-intervention, and follow-up to evaluate changes in adiposity.
  Units: Percentage (%)
Change in skeletal muscle mass, assessed by InBody 720 Bioimpedance Analyzer | From enrolment to 3 months after the intervention
  Skeletal muscle mass will be measured by the InBody 720 bioimpedance analyzer, providing an estimate of the muscle tissue mass in kilograms. Measurements at baseline, post-intervention, and follow-up will assess changes in muscle composition.
  Units: Kilograms (kg)
Change in Body Mass Index (BMI), calculated from InBody 720 measurements | From enrolment to 3 months after the intervention
  BMI will be calculated using the participant's weight and height measured or recorded during the study. BMI reflects the body mass relative to height squared (kg/m²). Changes in BMI will be assessed at baseline, post-intervention, and follow-up.
  Units: kg/m²
Change in visceral fat area, assessed by InBody 720 Bioimpedance Analyzer | From enrolment to 3 months after the intervention
  Visceral fat area, representing the fat surrounding internal organs, will be estimated by the InBody 720. Measurements at baseline, post-intervention, and follow-up will be used to monitor changes.
  Units: cm²
Baseline Self-Reported Physical Fitness (IFIS) vs. InBody 720 | At the baseline
  Self-reported physical fitness will be assessed at baseline using the International Fitness Scale (IFIS), a validated questionnaire measuring perceived fitness across five domains: general fitness, cardiorespiratory fitness, muscular strength, speed-agility, and flexibility. Each item is rated on a 5-point Likert scale from 1 (very poor) to 5 (very good). Higher scores indicate better perceived fitness. The total score is the mean or sum of item responses, depending on analysis strategy.
  Data will be collected digitally or on paper. Descriptive statistics and correlation analyses will be used to compare IFIS scores to objective measures from the InBody 720 bioimpedance analyzer, to assess alignment between subjective and objective fitness evaluations.
Assessed changes from baseline postural stability and balance control | From enrolment to 3 months after the intervention
  Balance and postural stability will be assessed using the BIODEX Stabilometric Platform. This device objectively measures static and dynamic balance, overall stability, and controlled mobility. Measurements will be taken at baseline, post-intervention, and follow-up to monitor changes in postural control and balance performance.
Assessed changes from baseline neuromuscular function (isokinetic dynamometry) | From enrolment to 3 months after the intervention
  Neuromuscular performance will be evaluated using the Biodex System 4 Pro, an advanced dynamometric system for assessing and training muscle function under various contraction modes. The device allows for testing in isometric, isotonic (concentric and eccentric), isokinetic (concentric and eccentric), reactive eccentric, and passive motion conditions. It provides objective data on muscle strength, endurance, and control, with full data archiving and export capabilities for statistical analysis. Measurements will be conducted at baseline, post-intervention, and follow-up to detect changes in neuromuscular function over time.
Assessed changes from baseline cardiopulmonary fitness (ergospirometry) | From enrolment to 3 months after the intervention
  Cardiopulmonary capacity will be evaluated using the Jaeger Oxycon Pro stationary ergospirometer, which analyzes exhaled gases during exercise to assess respiratory and circulatory function. The device uses precise O2 and CO2 analyzers to conduct Breath-by-Breath (3B) analysis, providing detailed functional assessments of the cardiovascular and pulmonary systems. Key parameters measured include maximum oxygen uptake (VO2 max), peak oxygen uptake (VO2 peak), ventilatory response to exercise (VE/VCO2 slope), and the respiratory exchange ratio (RER = VCO2/VO2), which is useful for evaluating anaerobic metabolism during exercise. These measurements will be taken at baseline, post-intervention, and follow-up to assess improvements in cardiorespiratory fitness.
Assessed changes from baseline lower limb power and force (vertical and horizontal jumping) | From enrolment to 3 months after the intervention
  Jumping ability and lower limb power will be assessed using the Kistler Model 9286BA dynamometric platform with MARS software. The platform, equipped with piezoelectric sensors, provides kinetic analysis of ground reaction forces during static and dynamic activities. It measures static body postural forces in a standing position, as well as dynamic forces during walking, running, and jumping. The platform captures both vertical and horizontal components of ground reaction forces during the support phase, enabling the evaluation of lower limb power, explosive strength, and maximal jump performance (e.g., vertical jump height and maximum power output). Measurements will be taken at baseline, post-intervention, and follow-up to assess changes in lower limb performance.
Assessed changes from baseline grip strength | From enrolment to 3 months after the intervention
  Grip strength will be measured using the SAEHAN electronic dynamometer with Herkules software. This device evaluates hand muscle strength by measuring grip force in an isometric test. The dynamometer features a five-level adjustable grip (ranging from 3.4 cm to 8.5 cm) to accommodate different hand sizes. The measurements will be taken at baseline, post-intervention, and follow-up to track changes in muscle strength and hand function.
Assessed changes from baseline blood lactate levels | From enrolment to the the end of the intervention
  Blood lactate concentration will be measured using the Lactate Scout 4 system. This device is designed for assessing lactate levels in capillary blood, providing insights into changes in physical fitness and endurance.
  Lactate levels will be measured by finger prick during the exercise test. A baseline assessment will be performed 5-7 minutes before the start of the test, then levels will be checked during the warm-up and twice during the exercise phase. Subsequent tests will be performed 2 and 5 minutes after the end of exercise. The test will be performed before the Onco-Move training intervention and after participation in 16 weeks of training (lactate levels tested seven times during each test).
Change in serum concentration of Interleukin-6 (IL-6) | From enrolment to 3 months after the intervention]
  IL-6 concentration will be measured in blood samples collected at baseline, post-intervention, and follow-up to assess inflammatory response. IL-6 is a pro-inflammatory cytokine associated with exercise-induced immune modulation.
  Units: pg/mL
Change in serum concentration of Interleukin-15 (IL-15) | From enrolment to 3 months after the intervention
  IL-15 will be measured to evaluate immune and metabolic responses to the intervention. This cytokine plays a role in skeletal muscle metabolism and immune signaling.
  Units: pg/mL
Change in serum concentration of Irisin | From enrolment to 3 months after the intervention
  Irisin levels will be assessed as a biomarker of exercise-induced metabolic activity and browning of adipose tissue.
  Units: ng/mL
Change in serum concentration of Brain-Derived Neurotrophic Factor (BDNF) | From enrolment to 3 months after the intervention
  BDNF will be measured to assess neuroplasticity and cognitive adaptations in response to the intervention. It is involved in neuronal survival, development, and synaptic plasticity.
  Units: ng/mL
Change in serum concentration of SPARC (Secreted Protein, Acidic and Rich in Cysteine) | From enrolment to 3 months after the intervention
  SPARC will be assessed to evaluate its role in exercise-induced muscle adaptation and extracellular matrix remodeling.
  Units: ng/mL
Change in serum concentration of Decorin | From enrolment to 3 months after the intervention
  Decorin will be analyzed as a marker of muscle regeneration and anti-fibrotic activity post-intervention.
  Units: ng/mL
Distribution of ACE Gene Polymorphisms | At the baseline
  Polymorphisms in the Angiotensin-Converting Enzyme (ACE) gene will be analyzed using blood samples to assess associations with cardiorespiratory and muscular adaptation to the intervention. Genotypes (e.g., I/I, I/D, D/D) will be reported.
  Unit of Measure: Proportion of participants with each genotype
Distribution of ACTN3 Gene Polymorphisms | At the baseline
  The ACTN3 polymorphism will be analyzed to explore associations with muscle strength and endurance performance.
  Unit of Measure: Proportion of participants with each genotype
Distribution of PPARGC1A Gene Polymorphisms | At the baseline
  Polymorphisms in the Peroxisome Proliferator-Activated Receptor Gamma Coactivator 1-alpha (PPARGC1A) gene will be examined for associations with mitochondrial function and metabolic adaptation.
Distribution of BDNF Gene Polymorphisms | At the baseline
  The BDNF Val66Met polymorphism will be genotyped to assess its role in neuroplasticity and mood changes in response to the intervention.
  Unit of Measure: Proportion of Val/Val, Val/Met, and Met/Met genotypes
Distribution of VEGF Gene Polymorphisms | At the baseline
  Polymorphisms in the VEGF gene will be analyzed to explore associations with vascular adaptation.
  Unit of Measure: Proportion of genotype variants
Distribution of IL6 Gene Polymorphisms | At the baseline
  The IL6 polymorphisms will be assessed for its role in inflammatory response to the intervention.
  Unit of Measure: Proportion of G/G, G/C, and C/C genotypes
Distribution of NOS3 Gene Polymorphisms | At the baseline
  NOS3 will be evaluated in relation to endothelial function and exercise response.
  Unit of Measure: Proportion of G/G, G/T, and T/T genotypes
Distribution of HIF1A Gene Polymorphisms | At the baseline
  HIF1A will be assessed for potential links with hypoxia tolerance and metabolic response.
  Unit of Measure: Proportion of Pro/Pro, Pro/Ser, and Ser/Ser genotypes
Distribution of TNF-α Gene Polymorphisms | At the baseline
  The TNF-α will be genotyped to examine inflammatory regulation. Unit of Measure: Proportion of G/G, G/A, and A/A genotypes
Distribution of mTOR Pathway Gene Polymorphisms | At the baseline
  Selected polymorphisms in genes from the mTOR pathway will be analyzed for associations with metabolic and muscular adaptation.
  Unit of Measure: Proportion of genotype variants
Change in relative telomere length and telomerase activity | From enrolment to 3 months after the intervention
  Telomere length and telomerase activity will be measured using qPCR or ELISA-based assays to evaluate cellular aging over the course of the intervention.
  Unit of Measure:
  * Telomere length: T/S ratio
  * Telomerase activity: Units per µg protein
Adherence to the mediterranean diet assessed by the 14-Item MEDAS Questionnaire | From Baseline up to 3 months after the intervention
  Adherence to a Mediterranean dietary pattern will be assessed using the 14-item Mediterranean Diet Adherence Screener (MEDAS), originally developed and validated in the PREDIMED trial. This questionnaire evaluates the frequency of consumption of key food components characteristic of the Mediterranean diet, such as olive oil, fruits, vegetables, legumes, nuts, fish, wine, and limits on red meat and processed foods. Each item is scored as 0 (does not meet the criterion) or 1 (meets the criterion), resulting in a total score ranging from 0 to 14, where higher scores indicate greater adherence to the Mediterranean diet.
  Unit of Measure: Score on a 0-14 scale

CONTACTS AND LOCATIONS:
Overall Officials: David Jiménez-Pavón, Professor, Study Director — Universidad de Cadiz
Locations (1):
- Gdansk University of Physical Education and Sport, Gdansk, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cufer T, Kosty MP; Curriculum Development Subgroup-ESMO/ASCO Global Curriculum Working Group. ESMO/ASCO Recommendations for a Global Curriculum in Medical Oncology Edition 2023. ESMO Open. 2023 Dec;8(6):101631. doi: 10.1016/j.esmoop.2023.101631. Epub 2023 Oct 23. PMID 38158226
- [Background] Vasilopoulou M, Asimakopoulou Z, Velissari J, Vicha A, Rizogianni M, Pusa S, Stoven S, Ficarra S, Bianco Alpha, Jimenez-Pavon D, Ponce Gonzalez Jesus G, Tavares Paula C, Gomes B, Bayer D, Silva S, Nogueira C, Papakonstantinou S, Musa K, Glorioso F, Vantarakis A. Interventions about physical activity and diet and their impact on adolescent and young adult cancer survivors: a Prisma systematic review. Support Care Cancer. 2024 May 13;32(6):342. doi: 10.1007/s00520-024-08516-0. PMID 38739198
- [Background] Ortega-Gomez S, Di Bartolo L, Velissari J, Gomes B, Pusa S, Thaller J, Papakonstantinou S, Kirkar M, Iannitto E, Moura N, Nogueira C, Ponce-Gonzalez JG, Baxter R, Tavares P, Vantarakis A, Bianco A, Carbonell-Baeza A, Jimenez-Pavon D; OACCUs consortium. Exploring the health benefits of outdoor exercise for cancer survivors: a systematic review of more than 700 individuals. Syst Rev. 2025 May 7;14(1):101. doi: 10.1186/s13643-025-02834-y. PMID 40336008
- [Background] Courneya KS, Vardy JL, O'Callaghan CJ, Gill S, Friedenreich CM, Wong RKS, Dhillon HM, Coyle V, Chua NS, Jonker DJ, Beale PJ, Haider K, Tang PA, Bonaventura T, Wong R, Lim HJ, Burge ME, Hubay S, Sanatani M, Campbell KL, Arthuso FZ, Turner J, Meyer RM, Brundage M, O'Brien P, Tu D, Booth CM; CHALLENGE Investigators. Structured Exercise after Adjuvant Chemotherapy for Colon Cancer. N Engl J Med. 2025 Jul 3;393(1):13-25. doi: 10.1056/NEJMoa2502760. Epub 2025 Jun 1. PMID 40450658
- [Background] Ng AH, Ngo-Huang A, Vidal M, Reyes-Garcia A, Liu DD, Williams JL, Fu JB, Yadav R, Bruera E. Exercise Barriers and Adherence to Recommendations in Patients With Cancer. JCO Oncol Pract. 2021 Jul;17(7):e972-e981. doi: 10.1200/OP.20.00625. Epub 2021 Mar 19. PMID 33739853
- [Background] Gunnell AS, Joyce S, Tomlin S, Taaffe DR, Cormie P, Newton RU, Joseph D, Spry N, Einarsdottir K, Galvao DA. Physical Activity and Survival among Long-term Cancer Survivor and Non-Cancer Cohorts. Front Public Health. 2017 Feb 14;5:19. doi: 10.3389/fpubh.2017.00019. eCollection 2017. PMID 28261579
- [Background] Felser S, Behrens M, Lampe H, Henze L, Grosse-Thie C, Murua Escobar H, Rohde K, Albrecht I, Zschorlich V, Junghanss C. Motivation and preferences of cancer patients to perform physical training. Eur J Cancer Care (Engl). 2020 Jul;29(4):e13246. doi: 10.1111/ecc.13246. Epub 2020 May 31. PMID 32476203
- [Background] Blaney JM, Lowe-Strong A, Rankin-Watt J, Campbell A, Gracey JH. Cancer survivors' exercise barriers, facilitators and preferences in the context of fatigue, quality of life and physical activity participation: a questionnaire-survey. Psychooncology. 2013 Jan;22(1):186-94. doi: 10.1002/pon.2072. Epub 2011 Oct 6. PMID 23296635
- [Background] Bray F, Laversanne M, Sung H, Ferlay J, Siegel RL, Soerjomataram I, Jemal A. Global cancer statistics 2022: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2024 May-Jun;74(3):229-263. doi: 10.3322/caac.21834. Epub 2024 Apr 4. PMID 38572751
- [Background] Miller KD, Fidler-Benaoudia M, Keegan TH, Hipp HS, Jemal A, Siegel RL. Cancer statistics for adolescents and young adults, 2020. CA Cancer J Clin. 2020 Nov;70(6):443-459. doi: 10.3322/caac.21637. Epub 2020 Sep 17. PMID 32940362
- [Background] Campbell KL, Winters-Stone KM, Wiskemann J, May AM, Schwartz AL, Courneya KS, Zucker DS, Matthews CE, Ligibel JA, Gerber LH, Morris GS, Patel AV, Hue TF, Perna FM, Schmitz KH. Exercise Guidelines for Cancer Survivors: Consensus Statement from International Multidisciplinary Roundtable. Med Sci Sports Exerc. 2019 Nov;51(11):2375-2390. doi: 10.1249/MSS.0000000000002116. PMID 31626055
- See also: Recruitment website — https://onkotrening.pl/onco-move/